CLINICAL TRIAL: NCT06227312
Title: Effect of Whole-body Vibration on the Ankle Joint, Plantar Pressure, and Running Paramethers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AWFiS/2023_6_PE
Record Dates: First submitted 2023-10-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-10

CONDITIONS: Range of Motion; Running; Gait
Keywords: runners; muscle flexibility; ankle; range of motion; foot arches; plantar pressure patterns; Footscan
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The participants engaged in four experimental sessions within 4 weeks. These sessions were conducted in a randomized sequence, with a one-week gap between each session. During each session, every participant performed one of the following tasks: 5 sets of 30 s calf raises on the platform but without vibration (CTRL); 5 sets of 30 s calf raises on the vibration platform with 30 s rest intervals between sets (WBV); 6 drop jump with a 30 s rest interval between sets (DJ); 5 sets of 30 s calf raises on the vibration platform followed by 6 drop jumps with a 30 s rest interval between sets (WBV + DJ).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- warm-up intervention (Experimental): Each participant performed all warm-up variants one week apart, without the possibility of repeating:
  CTRL 5 sets of 30 s calf raises on the platform but without vibration with 30 s rest intervals between sets; WBV 5 sets of 30 s calf raises on the vibration platform with 30 s rest intervals between sets; DJ 6 modified drop jump with a 30 s rest interval between sets (DJ); WBV + DJ 5 sets of 30 s calf raises on the vibration platform followed by 6 drop jumps with a 30 s rest interval between sets
  Interventions: Device: LADY 1 Pro, New Life Balance; Other: exercises

INTERVENTIONS:
Device: LADY 1 Pro, New Life Balance — whole-body vibration training on the platform
Other: exercises — calf raises and modified drop jumps

SUMMARY:
The main purpose of this study was the assessment of whole-body vibration warm-up, modified drop jumps, and combination of both on the range of motion of dorsiflexion in the ankle joint and running time. 16 recreationally active runners performed 4 different warm-up variants one week apart: 5 sets of 30 s calf raises on the platform but without vibration (CTRL), the same as CTRL group but with vibration with 30 s rest intervals between sets (WBV), 6 drop jumps with a 30 s rest interval between sets (DJ); last group was combination of both WBV and DJ groups (WBV+DJ). The study included muscle flexibility tests for the soleus and gastrocnemius muscles performed before the warm-up, 3 minutes after warm-up and immediately after a 3000 m run on a treadmill. The running time was measured and the run had to be completed in the shortest possible time.

Additionally, in the third week of the study there were performed static and dynamic foot measurements immediately before and after a 3000 m treadmill run. The main purpose of that gait analysis was to assess the impact of a 3km run on plantar pressure patterns and gait parameters in recreational runners.

ELIGIBILITY:
Inclusion Criteria:

* healthy and recreationally active males
* minimum two years of running training experience

Exclusion Criteria:

* rheumatological disease
* neurological disease
* orthopaedic disease
* genetic disease
* cardiovascular system disease
* pain in lower limbs in the last year
* pain in lumbar spine in the last year
* surgeries of lower limbs in the last year
* surgeries of spine in the last year
* musculoskeletal injuries in the lower limbs in the last year
* musculoskeletal injuries in the lumbar spine in the last year
* the absence during one or more training day

Ages: 34 Years to 42 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Ankle dorsiflexion range of motion (Gastrocnemius muscle flexibility test) | 3 times - before the warm-up, 3 minutes after warm-up and immediately after a 3000 m run
  The participant laid in a supine position with his knee straight and his ankle joint off the table. The researcher 1 tested the maximum dorsiflexion of the foot and controlled the position of the knee. The researcher 2 applied the AMI digital inclinometer (OPIW, Poland) to the outer edge of the foot. The The angle of dorsiflexion was measured in degrees.
Ankle dorsiflexion range of motion (Soleus muscle flexibility test) | 3 times - before the warm-up, 3 minutes after warm-up and immediately after a 3000 m run
  The participant laid in a supine position with the knee bent 90 degrees. The researcher 1 performed passive maximum dorsiflexion of the foot. The researcher 2 applied the AMI digital inclinometer (OPIW, Poland) to the outer edge of the foot. The angle of dorsiflexion was measured in degrees.
Static foot analysis (FootScan platform) | 2 times - immediately before and after 3000 m run
  In static measurement participants stood barefoot on the Footscan platform at a designated point, assuming a relaxed and natural position, remaining still and looking straight ahead with their arms by their sides. Static paramethers include the pressure of the parts of each foot (impulse - Ns/cm).
Dynamic foot analysis (FootScan platform) 1 | 2 times - immediately before and after 3000 m run
  During dynamic measurement participants were asked to walk barefoot in a relaxed manner at a self-selected comfort speed, and not to look at the ground. Dynamic parametrers include foot pressure (impulse - Ns/cm).
Dynamic foot analysis (FootScan platform) 2 | 2 times - immediately before and after 3000 m run
  During dynamic measurement participants were asked to walk barefoot in a relaxed manner at a self-selected comfort speed, and not to look at the ground. Dynamic parametrers include gait speed (m/s).
Dynamic foot analysis (FootScan platform) 3 | 2 times - immediately before and after 3000 m run
  During dynamic measurement participants were asked to walk barefoot in a relaxed manner at a self-selected comfort speed, and not to look at the ground. Dynamic parametrers include walking time (s).

CONTACTS AND LOCATIONS:
Overall Officials: Paulina W Ewertowska, PhD, Study Chair — Gdansk University of Physical Education and Sport
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Pomeranian Voivodeship, Poland